CLINICAL TRIAL: NCT06684327
Title: Multi-cohort, Single-arm Phase II Study of Albumin-paclitaxel, Ifosfamide, and Cisplatin in the Treatment of Rare Advanced Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, Director of oncologu department, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nab-TIP-001
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Paget Disease, Extramammary; Rhabdomyosarcoma; Testicular Cancer; Penile Cancer; Urachal Cancer
Keywords: rare tumor; albumin-paclitaxel; ifosfamide; cisplatin
MeSH Terms: conditions — Paget Disease, Extramammary; Rhabdomyosarcoma; Testicular Neoplasms; Penile Neoplasms; Urachal cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nab-TIP (Experimental): Participants will receive albumin-paclitaxel 260mg/m2 d1, isocyclophosphamide 1500mg/m2 d2-5, and cisplatin 25mg/m2 d2-5 every 21 days until disease progression, intolerable toxicity, or full 6 cycles of treatment, whichever occurs first.
  Interventions: Drug: Albumin-paclitaxel Injection

INTERVENTIONS:
Drug: Albumin-paclitaxel Injection — Participant will receive albumin-paclitaxel 260mg/m2 d1, isocyclophosphamide 1500mg/m2 d2-5, and cisplatin 25mg/m2 d2-5 every 21 days until disease progression, intolerable toxicity, or full 6 cycles of treatment, whichever occurs first.

SUMMARY:
The goal of this clinical trial is to learn if albumin-paclitaxel, ifosfamide and cisplatin (Nab-TIP) works to treat advanced rare tumors including PAGET's disease of scrotum with infiltrating sweat gland carcinoma （cohort 1）, rhabdomyosarcoma (cohort 2), testicular cancer (cohort 3), penile cancer (cohort 4), and urachus cancer (cohort 5) . It will also learn about the safety of Nab-TIP. The main questions it aims to answer are:

Does Nab-TIP improve the objective response rate and prolong the survival of participants? What medical problems do participants have when receiving the regimen of Nab-TIP?

Participants will:

Receive albumin-paclitaxel 260mg/m2 d1, isocyclophosphamide 1500mg/m2 d2-5, and cisplatin 25mg/m2 d2-5 every 21 days until disease progression, intolerable toxicity, or full 6 cycles of treatment, whichever occurs first.

Be performed imaging evaluation according to RECIST 1.1 every 6 weeks for 1 year of treatment and every 12 weeks after 1 year Be recorded any adverse events in the whole study period including type, incidence, grade, severity, duration, and association with the study drug according to NCI-CTCAE V5.0 criteria

DETAILED DESCRIPTION:
This study is a single-arm phase II study, which aimed to evaluate the efficacy and safety of albumin-paclitaxel, ifosfamide and cisplatin (Nab-TIP) in the treatment of advanced rare tumors including PAGET's disease of scrotum with infiltrating sweat gland carcinoma （cohort 1）, rhabdomyosarcoma (cohort 2), testicular cancer (cohort 3), penile cancer (cohort 4), and urachus cancer (cohort 5). Primary objective of this study is to evaluate the objective response rate (ORR) of Nab-TIP in the treatment of multiple rare advanced tumors. Secondary objectives are to evaluate the imaging progression-free survival (PFS), overall survival (OS) and safety in the treatment of multiple rare advanced tumors with Nab-TIP.

The study included a screening period (participants signed informed consent no more than 28 days before the first treatment in the study), a treatment period (treatment termination was defined as termination of treatment for any reason, such as imaging confirmation of disease progression, failure to tolerate adverse effects after dose adjustment, or early withdrawal for any reason), and a follow-up period (including end-of-treatment visits, safety visits, and survival follow-up).

Screening period: Participants are required to undergo a screening period within 28 days prior to the study's first treatment to determine eligibility.

Treatment period: Patients received albumin paclitaxel 260mg/m2 d1, isocyclophosphamide 1500mg/m2 d2-5, cisplatin 25mg d2-5, repeated every three weeks, with 6 cycles of chemotherapy.

Follow-up period: The safety follow-up period began after the last study treatment, and was followed up once on the 30th day (±7 days). Subjects should go to the research center for the examination of vital signs, physical examination, laboratory examination and other protocol requirements, and evaluate AE, concomitant medication and concomitant treatment.

After the end of the safety follow-up period, the subjects entered the 1-year survival follow-up period, which was conducted every 3 months. They could be visited by telephone follow-up and other effective ways to collect survival information and follow-up treatment information. Survival follow-up lasted until death, loss of follow-up, withdrawal of informed consent, or investigator termination of the study

ELIGIBILITY:
Inclusion Criteria:

* Individuals able to understand and give written informed consent.
* Histologically or cytologically confirmed cancer of one of the following types:

PAGET's disease of scrotum with infiltrating sweat gland carcinoma Rhabdomyosarcoma Testicular cancer Penile cancer Urachal cancer

* Stage IV disease
* Adequate performance status (ECOG 0-2)
* Expected survival ≥ 3 months.
* Measurable disease by CT or MRI, Or lesions with skin infiltration.
* Adequate hematology without ongoing transfusional support (hemoglobin > 9 g/dL, absolute neutrophil count (ANC) > 1,500 per mm^3, platelets > 100,000 per mm^3).
* Adequate renal and hepatic function (creatinine ≤ 2.0 x institutional upper limit of normal (IULN), bilirubin ≤ 1.5 IULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x IULN or 5 x IULN if know liver metastases).
* Adequate coagulation function: International Normalized Ratio (INR) ≤1.5 /PT≤1.5×ULN, aPTT≤1.5×ULN.
* Willing to use a medically approved contraceptive method from the enrollment to at least 120 days after the end of the study, and sperm donation to another person or cryopreservation for fertilization and reproduction is not permitted during this period.
* Ability to comply with research visit schedules and other protocol requirements.

Exclusion Criteria:

* 1. Active or uncontrolled severe infections (≥CTCAE Level 2) requiring systemic antibacterial, antifungal, or antiviral therapy, including tuberculosis infections.
* 2. Active hepatitis (transaminases not within inclusion criteria; HBV reference: HBV DNA ≥2000 IU/ml or ≥10^4 copies/ml; HCV reference: HCV RNA ≥2000 IU/ml or ≥10^4 copies/ml; after nucleoside antiviral treatment below the above standards, may be eligible; chronic HBV carrier with HBV DNA <10^4 IU/ml, must receive antiviral treatment during the study period to be eligible).
* 3. Renal failure requiring hemodialysis or peritoneal dialysis.
* 4. History of immunodeficiency, including HIV positive or having other acquired/congenital immunodeficiency diseases, or organ transplant history.
* 5. Severe nausea, headache, insomnia, fatigue, somnolence, dry mouth, dizziness, and constipation.
* 6. History of active tuberculosis.
* 7. Uncontrolled ascites, pleural effusion, or pericardial effusion requiring repeated drainage.
* 8. Patients who have undergone major organ transplantation.
* 9. Individuals who have undergone major surgical procedures, open biopsies, or obvious traumatic injuries within 28 days prior to the start of the study; or have unhealed wounds or fractures for a long time;
* 10. Individuals who have participated or are currently participating in another clinical study within the past 4 weeks prior to the start of the study;
* 11. Individuals with a history of severe allergies;
* 12. Individuals at risk of bleeding, or with impaired coagulation function, or who are currently receiving thrombolytic therapy;
* 13. Individuals with a history of substance abuse with no ability to abstain or with a mental disorder.
* 14. According to the investigator's judgment, subjects with serious adverse effects on their safety or completion of the study, or those with accompanying diseases that seriously endanger the safety of the subjects or affect the completion of the study, or those with other reasons deemed unsuitable for enrollment by the investigator. Subjects with a history of a clearly defined neurological or psychiatric disorder, such as dementia, epilepsy, or a history of epilepsy prone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 weeks
  ORR was defined as the proportion of patients who achieved either a complete response (CR) or a partial response (PR) based on the investigator's assessment (RECIST v1.1) that was confirmed by a subsequent scan ≥4 weeks after initial CR/PR.

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 1 year
  PFS was defined as the time between the enrollment and either RECIST1.1-defined progressive disease or death due to any cause, whichever occurred first.
Overall survival (OS) | 2 years
  OS was defined as the time between the enrollment and death due to any cause.

OTHER OUTCOMES:
Adverse events (AE) | 2 years
  Any adverse events will be recorded in the whole study period including type, incidence, grade, severity, duration, and association with the study drug according to NCI-CTCAE V5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Wang, Doctor, Study Director — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No